CLINICAL TRIAL: NCT03447899
Title: Longitudinal, Multi-Dimensional Assessment of Recovery and Added Benefit of a Behavioral Health Intervention for Children With Abusive Head Trauma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-1221; IHEA101376 (Other Grant/Funding Number: Colorado Department of Human Services)
Record Dates: First submitted 2018-01-10; First posted 2018-02-27 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Non-Accidental Traumatic Head Injury to Child

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABC Intervention (Experimental): The investigators will deliver the "Attachment and Biobehavioral Catch-up (ABC)" in the home weekly using live, in-room coaching, to give caregivers feedback as they use targeted skills during interactions with the child. The intervention will last 10 sessions. Study participants in both groups will complete study measures at baseline, 1 month, 3 months, post-intervention, 6 months, and 12 months.
  Interventions: Behavioral: Attachment and Biobehavioral Catch-up (ABC)
- Standard of Care (No Intervention): Subjects will receive normal standard of care without the "Attachment and Biobehavioral Catch-up (ABC)".

INTERVENTIONS:
Behavioral: Attachment and Biobehavioral Catch-up (ABC) — Attachment and Biobehavioral Catch-up (ABC) is an in-home, 10-session, manualized parent-training program for children ages 6 months through 2 years who have experienced early adversity. ABC utilizes parent-child interactions to enhance positive interactions with the child through live coaching with particular focus on nurturing behaviors, following the child's lead, non-frightening behaviors. These behaviors include appropriate soothing and comforting when a child is distressed, responding to or imitating a child in a contingent way, and displaying warmth.
  Arms: ABC Intervention

SUMMARY:
Family dynamics and caregiver responses to a child with traumatic brain injury are implicated both as precipitating events as well as factors influencing outcomes of abusive head trauma (AHT). However, no family behavioral health intervention exists to meet the unique needs of families with infants and very young children with AHT. The study was initially designed as a randomized controlled trial (RCT) to assess the efficacy of an evidence-based behavioral intervention to improve outcomes for families and children with AHT. However, rates of recruitment were so low that the investigators and funder amended the study to be intervention only (with IRB approval). At that time, there were five participants and only one had been assigned to the intervention arm. Only one additional family was recruited, and that family did not complete study measures prior to the time at which the intervention would start and did not receive the intervention. The investigators did examine outcomes in multiple dimensions, including clinical, cognitive, family, caregiver, child behavior, and service usage over time but connot compare to patients not receiving the intervention. The investigators were not able to examine characteristics of patients and families best suited for this behavioral health intervention.

DETAILED DESCRIPTION:
27 children (ages 3 months to 2 years) and their caregiver referred to the Non-Accidental Brain Injury Care Clinic at the Children's Hospital Colorado (CHCO) were recruited for participation in the study, 7 families consented. One family received the Attachment and Biobehavioral (ABC) intervention. One family discontinued participation. The data collection schedule was 1 month post-injury, 3 months, 6 months, 9 months, and 12 months. Outcomes in multiple dimensions, were assessed including clinical recovery, cognitive, language, and motor functioning, family functioning, caregiver mental health including anxiety, depression, competency, and stress. The investigators also examined service use over time. Analyses will assess trajectories of recovery for both groups using data for all time points.

ELIGIBILITY:
Inclusion Criteria:

* Children who have experienced AHT as determined by the CHCO Child Protection Team
* Caregivers who speak English
* Families who live in the Denver Metro area and,
* Child-victim age between 3 months and 2 years of age

Exclusion Criteria:

* Those with significant disability that would inhibit participation in the intervention,
* Those scoring below 6 months on developmental measures will not be eligible.

Ages: 3 Months to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 7 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of cognitive scores of children receiving the ABC intervention to those receiving usual care. | 6 months
  Compare the Cognitive scale standard score from the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The cognitive scale standard score ranges from 50-150. Higher scores indicate better cognitive functioning.
Evaluation of motor scores of children receiving the ABC intervention to those receiving usual care. | 6 months
  Compare the overall Motor standard score from the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The overall Motor score is a combined score from the Gross Motor and Fine Motor Scales of the Bayley III. The overall motor score is a summed value from the Gross Motor and Fine Motor subscales. Subscale scores are added, then standardized (Mean = 100, SD =15). The range of values for the overall Motor standard score is 50-150. Higher values indicate better motor functioning.
Evaluation of socioemotional scores of children receiving the ABC intervention to those receiving care as usual. | 6 months
  Compare scores from the Social-Emotional standard score on the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The range of values for the Social-Emotional Scale is 50-150. Higher values indicate better social-emotional functioning.
Evaluation of language scores of children receiving the ABC intervention to those receiving care as usual. | 6 months
  Compare scores on the overall language score on the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The overall language score is the summed score from the Expressive Language and Receptive Language subscales. The summed value is then standardized (mean = 100, SD = 15). The range of values are 50-150. Higher values indicate better language functioning.
Evaluation of depression scores of caregivers receiving the ABC intervention to those receiving care as usual. | 6 months
  Compare caregiver depression scores of those receiving the intervention to those receiving care as usual. Depression is measured using the Center for Epidemiological Depression Scale (CES-D). Values range from 0-60. Higher values indicate greater depressive symptoms.
Evaluation of anxiety scores of caregivers receiving the ABC intervention to those receiving care as usual. | 6 months
  Compare caregiver scores from the Generalized Anxiety scale (GAD) of those receiving the intervention to those receiving care as usual. The range of values is 0 -21. Higher values indicate greater anxiety symptoms.
Evaluation of parenting stress scores of caregivers receiving the ABC intervention to those receiving care as usual. | 6 months
  Compare scores on the Parenting Stress Index-Short Form of those receiving the intervention to those receiving care as usual. Scores on the PSI-SF are a sum of scores from non-duplicate items from the Parental Distress subscale, Parent-child dysfunctional interaction subscale, and the difficult child subscale. Range of values for the total score are 36-180. Higher values indicate greater parental distress.
Evaluation of family functioning of caregivers receiving the ABC intervention to those receiving care as usual. | 6 months
  Compare scores from the General Functioning subscale of the Family Assessment Device of those receiving the intervention to those receiving care as usual. Scores on the General Functioning subscale range from 12 to 48. Higher values indicate greater family dysfunction.
Evaluation of screener scores of child abuse risk of caregivers receiving the ABC intervention to those receiving care as usual. | 6 months
  Compare scores on the Child Abuse Potential Inventory -Brief Version of caregivers receiving the intervention to those receiving care as usual. Scores on the brief version range from 0-34. Higher scores indicate greater potential risk of child abuse.
Evaluation of caregiver reported service utilization for children receiving the ABC intervention to those receiving care as usual. | 6 months
  Compare the utilization of occupational, physical, speech, vision, feeding, or developmental therapy, as well as receipt of nursing care and family psychological services of those families receiving the intervention compared to those receiving care as usual. Service utilization is captured through a project developed measure asking the respondent if his/her child received any service on the list of services since the last interview period. Any endorsement of any service will be coded affirmative. Indicators of use of those receiving the intervention will be compare to those receiving care as usual.
Evaluation of cognitive scores of children receiving the ABC intervention to those receiving usual care. | 9 months
  Compare the Cognitive scale standard score from the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The cognitive scale standard score ranges from 50-150. Higher scores indicate better cognitive functioning.
Evaluation of cognitive scores of children receiving the ABC intervention to those receiving usual care. | 12 months
  Compare the Cognitive scale standard score from the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The cognitive scale standard score ranges from 50-150. Higher scores indicate better cognitive functioning.
Evaluation of motor scores of children receiving the ABC intervention to those receiving usual care. | 9 months
  Compare the overall Motor standard score from the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The overall Motor score is a combined score from the Gross Motor and Fine Motor Scales of the Bayley III. The overall motor score is a summed value from the Gross Motor and Fine Motor subscales. Subscale scores are added, then standardized (Mean = 100, SD =15). The range of values for the overall Motor standard score is 50-150. Higher values indicate better motor functioning.
Evaluation of motor scores of children receiving the ABC intervention to those receiving usual care. | 12 months
  Compare the overall Motor standard score from the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The overall Motor score is a combined score from the Gross Motor and Fine Motor Scales of the Bayley III. The overall motor score is a summed value from the Gross Motor and Fine Motor subscales. Subscale scores are added, then standardized (Mean = 100, SD =15). The range of values for the overall Motor standard score is 50-150. Higher values indicate better motor functioning.
Evaluation of socioemotional scores of children receiving the ABC intervention to those receiving care as usual. | 9 months
  Compare scores from the Social-Emotional standard score on the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The range of values for the Social-Emotional Scale is 50-150. Higher values indicate better social-emotional functioning.
Evaluation of socioemotional scores of children receiving the ABC intervention to those receiving care as usual. | 12 months
  Compare scores from the Social-Emotional standard score on the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The range of values for the Social-Emotional Scale is 50-150. Higher values indicate better social-emotional functioning.
Evaluation of language scores of children receiving the ABC intervention to those receiving care as usual. | 9 months
  Compare scores on the overall language score on the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The overall language score is the summed score from the Expressive Language and Receptive Language subscales. The summed value is then standardized (mean = 100, SD = 15). The range of values are 50-150. Higher values indicate better language functioning.
Evaluation of language scores of children receiving the ABC intervention to those receiving care as usual. | 12 months
  Compare scores on the overall language score on the Bayley Scales of Infant and Toddler Development-Third Edition of those receiving the intervention to those receiving care as usual. The overall language score is the summed score from the Expressive Language and Receptive Language subscales. The summed value is then standardized (mean = 100, SD = 15). The range of values are 50-150. Higher values indicate better language functioning.
Evaluation of depression scores of caregivers receiving the ABC intervention to those receiving care as usual. | 9 months
  Compare caregiver depression scores of those receiving the intervention to those receiving care as usual. Depression is measured using the Center for Epidemiological Depression Scale (CES-D). Values range from 0-60. Higher values indicate greater depressive symptoms.
Evaluation of depression scores of caregivers receiving the ABC intervention to those receiving care as usual. | 12 months
  Compare caregiver depression scores of those receiving the intervention to those receiving care as usual. Depression is measured using the Center for Epidemiological Depression Scale (CES-D). Values range from 0-60. Higher values indicate greater depressive symptoms.
Evaluation of anxiety scores of caregivers receiving the ABC intervention to those receiving care as usual. | 9 months
  Compare caregiver scores from the Generalized Anxiety scale (GAD) of those receiving the intervention to those receiving care as usual. The range of values is 0 -21. Higher values indicate greater anxiety symptoms.
Evaluation of anxiety scores of caregivers receiving the ABC intervention to those receiving care as usual. | 12 months
  Compare caregiver scores from the Generalized Anxiety scale (GAD) of those receiving the intervention to those receiving care as usual. The range of values is 0 -21. Higher values indicate greater anxiety symptoms.
Evaluation of parenting stress scores of caregivers receiving the ABC intervention to those receiving care as usual. | 9 months
  Compare scores on the Parenting Stress Index-Short Form of those receiving the intervention to those receiving care as usual. Scores on the PSI-SF are a sum of scores from non-duplicate items from the Parental Distress subscale, Parent-child dysfunctional interaction subscale, and the difficult child subscale. Range of values for the total score are 36-180. Higher values indicate greater parental distress.
Evaluation of parenting stress scores of caregivers receiving the ABC intervention to those receiving care as usual. | 12 months
  Compare scores on the Parenting Stress Index-Short Form of those receiving the intervention to those receiving care as usual. Scores on the PSI-SF are a sum of scores from non-duplicate items from the Parental Distress subscale, Parent-child dysfunctional interaction subscale, and the difficult child subscale. Range of values for the total score are 36-180. Higher values indicate greater parental distress.
Evaluation of family functioning of caregivers receiving the ABC intervention to those receiving care as usual. | 9 months
  Compare scores from the General Functioning subscale of the Family Assessment Device of those receiving the intervention to those receiving care as usual. Scores on the General Functioning subscale range from 12 to 48. Higher values indicate greater family dysfunction.
Evaluation of family functioning of caregivers receiving the ABC intervention to those receiving care as usual. | 12 months
  Compare scores from the General Functioning subscale of the Family Assessment Device of those receiving the intervention to those receiving care as usual. Scores on the General Functioning subscale range from 12 to 48. Higher values indicate greater family dysfunction.
Evaluation of screener scores of child abuse risk of caregivers receiving the ABC intervention to those receiving care as usual. | 9 months
  Compare scores on the Child Abuse Potential Inventory -Brief Version of caregivers receiving the intervention to those receiving care as usual. Scores on the brief version range from 0-34. Higher scores indicate greater potential risk of child abuse.
Evaluation of screener scores of child abuse risk of caregivers receiving the ABC intervention to those receiving care as usual. | 12 months
  Compare scores on the Child Abuse Potential Inventory -Brief Version of caregivers receiving the intervention to those receiving care as usual. Scores on the brief version range from 0-34. Higher scores indicate greater potential risk of child abuse.
Evaluation of caregiver reported service utilization for children receiving the ABC intervention to those receiving care as usual. | 9 months
  Compare the utilization of occupational, physical, speech, vision, feeding, or developmental therapy, as well as receipt of nursing care and family psychological services of those families receiving the intervention compared to those receiving care as usual. Service utilization is captured through a project developed measure asking the respondent if his/her child received any service on the list of services since the last interview period. Any endorsement of any service will be coded affirmative. Indicators of use of those receiving the intervention will be compare to those receiving care as usual.
Evaluation of caregiver reported service utilization for children receiving the ABC intervention to those receiving care as usual. | 12 months
  Compare the utilization of occupational, physical, speech, vision, feeding, or developmental therapy, as well as receipt of nursing care and family psychological services of those families receiving the intervention compared to those receiving care as usual. Service utilization is captured through a project developed measure asking the respondent if his/her child received any service on the list of services since the last interview period. Any endorsement of any service will be coded affirmative. Indicators of use of those receiving the intervention will be compare to those receiving care as usual.

SECONDARY OUTCOMES:
Evaluation clusters of patient and family characteristics that benefit most from a parenting intervention component | 1 month, 3 month, 6 months, 9 months, 12 months
  Compare any changes in Demographic, family, and injury data aggregated in a latent class approach to identify which constellations of risk and protective factors were most amenable to the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Terri H Lewis, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Children's Hospital of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No